CLINICAL TRIAL: NCT05107583
Title: Comparing the Effects of a High- and Low-carbohydrate Pre-exercise Meal Relative to Fasting on Exercise Metabolism, Subsequent Appetite, and Energy Intake in Healthy Males.
Brief Title: Effects of Pre-exercise Carbohydrate Restriction Relative to Fasting on Metabolism, Appetite, and Energy Intake in Healthy Males.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham Trent University (Other)
Collaborators: Loughborough University (Other)
Responsible Party: Principal Investigator, Tommy Slater, Principle Investigator, Nottingham Trent University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: TS_PreExCHO_2021
Record Dates: First submitted 2021-08-12; First posted 2021-11-04 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Obesity; Metabolic Syndrome
Keywords: Fasted exercise; Low-carbohydrate; High-protein; Appetite; Energy Intake; Metabolism
MeSH Terms: conditions — Obesity; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: The study design is a randomised, controlled, crossover design in which participants undertake three exercise conditions in a randomised order with at least a seven day period in between trials.
Who Masked: Participant
Masking Description: Due to the obvious differences between fasting and consuming food, participants will be aware of when they have been assigned to the fasted condition. However, the low- and high-carbohydrate content lunch meals will be closely matched for taste, with carbohydrate content being manipulated within a drink. Participants will not be informed that the carbohydrate content of the lunch meals is being manipulated, and will therefore, be blinded to this element of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-Carbohydrate Pre-Exercise Meal (Experimental): Participants will consume a low-carbohydrate (<10% carbohydrate) lunch meal at 13:30 - 2.5 hours prior to commencing exercise at 16:00.
  Interventions: Behavioral: Low-Carbohydrate Pre-Exercise Meal
- High-Carbohydrate Pre-Exercise Meal (Experimental): Participants will consume a high-carbohydrate (~2.2 g/kg carbohydrate) lunch meal at 13:30 - 2.5 hours prior to commencing exercise at 16:00.
  Interventions: Behavioral: High-Carbohydrate Pre-Exercise Meal
- Fasted Exercise (Experimental): Participants will skip lunch, and continue fasting since breakfast (08:00) before commencing exercise at 16:00. Therefore, exercise will commence after an 8 hour period of fasting.
  Interventions: Behavioral: Fasted Exercise

INTERVENTIONS:
Behavioral: Low-Carbohydrate Pre-Exercise Meal — Sixty minutes of cycling at 60% VO2peak will take place on a stationary bicycle ergometer at 16:00, after having consumed a low-carbohydrate lunch meal (<10% carbohydrate; 35% estimated energy requirements) 2.5 hours prior.
  Arms: Low-Carbohydrate Pre-Exercise Meal
Behavioral: High-Carbohydrate Pre-Exercise Meal — Sixty minutes of cycling at 60% VO2peak will take place on a stationary bicycle ergometer at 16:00, after having consumed a high-carbohydrate lunch meal (~2.2 g/kg carbohydrate; 35% estimated energy requirements) 2.5 hours prior.
  Arms: High-Carbohydrate Pre-Exercise Meal
Behavioral: Fasted Exercise — Sixty minutes of cycling at 60% VO2peak will take place on a stationary bicycle ergometer at 16:00, after having skipped lunch, and having consumed nothing other than plain water since breakfast (08:00; 25% estimated energy requirements). Exercise will therefore commence after an 8 hour period of fasting.
  Arms: Fasted Exercise

SUMMARY:
This study will compare the metabolic, appetite, energy intake, and perceptual responses to a bout of exercise completed in the evening after after a low-carbohydrate lunch meal (<10% carbohydrate content / 0.2 g/kg carbohydrate; LO-CHO), with the responses to exercise performed after a lunch meal containing a high carbohydrate content (~60% carbohydrate content / 2.2 g/kg carbohydrate; HI-CHO), and after skipping lunch and fasting for 8 hours since breakfast (FAST).

DETAILED DESCRIPTION:
Regular exercise is known to be a successful strategy for improving several facets of health and maintaining body weight. However, many people are not engaging in enough exercise, and some may not be achieving maximum benefits from the exercise that they already do. Performing exercise in the overnight fasted state has been shown to reduce energy intake over the course of a single day, without any compensatory reductions in free-living energy expenditure. Despite these promising findings, it is likely that not every member of the population is logistically able to perform exercise in the morning due to various work, family and social commitments, and exercise in the evening may be a logical alternative for these individuals.

Studies have found that exercise performed after an overnight fast may incur superior improvements in insulin sensitivity in lean individuals (Van Proeyen et al., 2010), and individuals with overweight or obesity (Edinburgh et al., 2020), compared to exercising after breakfast. These superior improvements may be mediated, in part, by an increased mobilisation and oxidation of endogenous lipid stores. Additionally, overnight fasted exercise may result in a more negative energy balance than exercising after breakfast (Bachman et al., 2016; Edinburgh et al., 2019). We recently examined whether exercise performed in the evening following an extended period of fasting (7 h) would induce similar responses to overnight fasted exercise regarding substrate oxidation patterns and subsequent energy intake (manuscript in preparation - NCT04742530). This research question was important, as we speculate that a large proportion of the population are likely unable to perform exercise in the morning after an overnight fast due to various logistical barriers. Therefore fasting prior to evening exercise could act as an alternative for these individuals.

We found that compared to consuming a carbohydrate-containing meal 2 h prior, fasting before evening exercise resulted in elevated fat oxidation rates during exercise, but was accompanied by compensatory eating at dinner. Additionally, participants reported that fasting throughout the afternoon was difficult. The long-term efficacy of fasted evening exercise may, therefore, be limited by increased hunger and compensatory energy intake.

Consuming a meal lower in carbohydrate and higher in protein and/or fat can increase rates of fat oxidation during exercise (Rowlands & Hopkins, 2002; Oliviera et al., 2021). Protein is also the most satiating macronutrient, and high-protein diets are associated with reductions in energy intake. Consuming a high-protein pre-exercise meal compared to a typical high-carbohydrate meal also led to greater exercise-induced elevations in hormones typically associated with increased satiety and reduced hunger: peptide tyrosine-tyrosine (PYY) and glucagon-like peptide-1 (GLP-1) (Oliviera et al., 2021). Therefore, consuming a meal with a low carbohydrate content and higher protein content before exercise, rather than completely fasting, could be utilised to enhance the metabolic responses to exercise, whilst simultaneously managing appetite and subsequent energy intake. Further research is needed to fully understand the metabolic and appetite-related effects of a low-carbohydrate, higher-protein meal prior to exercise in the evening, compared to a typically consumed higher-carbohydrate meal and complete fasting.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smokers (due to the well-known impact of smoking on appetite.
2. Not currently on a weight management program or have an unusual eating pattern (i.e., extended fasting periods >8 h other than overnight).
3. Have maintained a stable weight for 6 months (self-reported).
4. No history of gastric, digestive, cardiovascular or renal disease (self-reported).

Exclusion Criteria:

1. Severe food allergies, dislike or intolerance of study foods or drinks.
2. Currently undergoing a lifestyle intervention (structured diet or exercise).
3. Diagnosis of a condition or currently undergoing treatment therapy known to affect glucose or lipid metabolism (e.g., type-2 diabetes, taking statins), or contraindications to exercise.
4. Use of medication or supplements that may affect hormone concentrations and/or substrate metabolism.
5. Excessive alcohol consumption (>14 units/week).
6. Intensive training schedule (>10 hours/week).

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Fat Oxidation Rate During Steady-State Exercise. | Throughout the 60-minute steady-state bout of cycling
  Measurements of VO2 and VCO2 during a 60 minute steady state bout of cycling to determine rates of fat oxidation.

SECONDARY OUTCOMES:
Voluntary energy intake (Kilocalories) at a laboratory-based test meal. | 60 minutes following the end of the exercise session.
  A laboratory-based dinner meal consisting of pasta, tomato sauce and olive oil will be provided to participants in excess of expected consumption. Participants will be permitted 20 minutes to eat as much or as little as they desire, until 'comfortably full and satisfied'.
Visual Analogue Scale for Subjective Ratings of Appetite. | Baseline, 1 hour, 1.75 hours, 2.75 hours, 3 hours, 3.5 hours (mid-exercise), 4 hours, 5 hours.
  Time-course of subjective ratings of hunger between breakfast provision and one hour after consuming lunch, measured using an appetite visual analogue scale. The scale is divided into subscales of different appetite perceptions including: hunger, fullness, desire to eat and prospective food consumption. Each subscale is rated on a 100mm scale (i.e. from 0 - 100), with a rating of 100 fully supporting the perception and a rating of 0 fully opposing the perception.
Acylated ghrelin | Baseline, 1 hour, 1.75 hours, 2.75 hours, 3 hours, 3.5 hours (mid-exercise), 4 hours, 5 hours.
  Time-course of acylated ghrelin plasma concentrations across experimental trials.
Peptide tyrosine-tyrosine (PYY) | Baseline, 1 hour, 1.75 hours, 2.75 hours, 3 hours, 3.5 hours (mid-exercise), 4 hours, 5 hours.
  Time-course of PYY plasma concentrations across experimental trials.
Glucagon-like peptide-1 (GLP-1) | Baseline, 1 hour, 1.75 hours, 2.75 hours, 3 hours, 3.5 hours (mid-exercise), 4 hours, 5 hours.
  Time-course of GLP-1 plasma concentrations across experimental trials.
Glucose | Baseline, 1 hour, 1.75 hours, 2.75 hours, 3 hours, 3.5 hours (mid-exercise), 4 hours, 5 hours.
  Time-course of glucose plasma concentrations across experimental trials.
Insulin | Baseline, 1 hour, 1.75 hours, 2.75 hours, 3 hours, 3.5 hours (mid-exercise), 4 hours, 5 hours.
  Time-course of insulin plasma concentrations across experimental trials.
Non-esterified fatty-acids (NEFA) | Baseline, 1 hour, 1.75 hours, 2.75 hours, 3 hours, 3.5 hours (mid-exercise), 4 hours, 5 hours.
  Time-course of NEFA plasma concentrations across experimental trials.
Glycerol | Baseline, 1 hour, 1.75 hours, 2.75 hours, 3 hours, 3.5 hours (mid-exercise), 4 hours, 5 hours.
  Time-course of glycerol plasma concentrations across experimental trials.
Rating of Perceived Exertion (RPE). | Throughout the 60-minute steady-state bout of cycling.
  RPE will be measured at 10-minute intervals throughout the 60-minute exercise period on a 6-20 RPE scale. The participant will point to the value that corresponds to their current perceived exertion (6 being no exertion at all; 20 being maximal exertion).
Pre-exercise Subjective Feelings. | Immediately before the exercise session.
  A single questionnaire to assess pre-exercise subjective feelings will be measured using a visual analogue scale. The scale is divided into subscales of different feelings including: motivation, readiness, tiredness, nausea, and energetic. Each subscale is rated on a 100mm scale (i.e. from 0 - 100), with a rating of 100 fully supporting the perception and a rating of 0 fully opposing the perception.
Enjoyment of the Exercise Bout. | Immediately following the end of the exercise session.
  A shortened version of The Physical Activity Enjoyment Scale (PACES) will be completed to gauge enjoyment of the exercise sessions. A scale from 1-7 will be used for eight feelings. The participant will circle the value that corresponds to which (6 being no exertion at all; 20 being maximal exertion).
  The scale is divided into bipolar subscales of different feelings including: enjoyment, liking, pleasure, fun, pleasantness, interest, engagement and task absorption . Each subscale is rated on a 1-7 bipolar scale (i.e. from 1 - 7), with a rating of 1 fully supporting the feeling on the left-hand side of the subscale, and a rating of 7 fully supporting the feeling on the right-hand side of the subscale. For three subscales, a positive feeling is placed at 7, and for four subscales, a negative feeling is placed at 7 (reverse scored).
Carbohydrate Oxidation Rate During Steady-State Exercise | Throughout the 60-minute steady-state bout of cycling
  Measurements of VO2 and VCO2 during a 60 minute steady state bout of cycling to determine rates of carbohydrate oxidation
Rate of Energy Expenditure During Steady-State Exercise | Throughout the 60-minute steady-state bout of cycling
  Measurements of VO2 and VCO2 during a 60 minute steady state bout of cycling to determine rates energy expenditure.
Carbohydrate Oxidation Rate At Rest | Baseline, 1 hour, 1.75 hours, 2.75 hours, 5 hours
  Measurements of VO2 and VCO2 during at rest during experimental trials to determine rates of carbohydrate oxidation.
Fat Oxidation Rate At Rest | Baseline, 1 hour, 1.75 hours, 2.75 hours, 5 hours
  Measurements of VO2 and VCO2 during at rest during experimental trials to determine rates of fat oxidation.
Rate of Energy Expenditure At Rest | Baseline, 1 hour, 1.75 hours, 2.75 hours, 5 hours
  Measurements of VO2 and VCO2 during at rest during experimental trials to determine rates of energy expenditure.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Loughborough University, Loughborough, Leicestershire
  - Nottingham Trent University, Nottingham, Nottinghamshire

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Edinburgh RM, Bradley HE, Abdullah NF, Robinson SL, Chrzanowski-Smith OJ, Walhin JP, Joanisse S, Manolopoulos KN, Philp A, Hengist A, Chabowski A, Brodsky FM, Koumanov F, Betts JA, Thompson D, Wallis GA, Gonzalez JT. Lipid Metabolism Links Nutrient-Exercise Timing to Insulin Sensitivity in Men Classified as Overweight or Obese. J Clin Endocrinol Metab. 2020 Mar 1;105(3):660-76. doi: 10.1210/clinem/dgz104. PMID 31628477
- [Background] Van Proeyen K, Szlufcik K, Nielens H, Pelgrim K, Deldicque L, Hesselink M, Van Veldhoven PP, Hespel P. Training in the fasted state improves glucose tolerance during fat-rich diet. J Physiol. 2010 Nov 1;588(Pt 21):4289-302. doi: 10.1113/jphysiol.2010.196493. PMID 20837645
- [Background] Edinburgh RM, Hengist A, Smith HA, Travers RL, Betts JA, Thompson D, Walhin JP, Wallis GA, Hamilton DL, Stevenson EJ, Tipton KD, Gonzalez JT. Skipping Breakfast Before Exercise Creates a More Negative 24-hour Energy Balance: A Randomized Controlled Trial in Healthy Physically Active Young Men. J Nutr. 2019 Aug 1;149(8):1326-1334. doi: 10.1093/jn/nxz018. PMID 31321428
- [Background] Bachman JL, Deitrick RW, Hillman AR. Exercising in the Fasted State Reduced 24-Hour Energy Intake in Active Male Adults. J Nutr Metab. 2016;2016:1984198. doi: 10.1155/2016/1984198. Epub 2016 Sep 21. PMID 27738523
- [Background] Rowlands DS, Hopkins WG. Effects of high-fat and high-carbohydrate diets on metabolism and performance in cycling. Metabolism. 2002 Jun;51(6):678-90. doi: 10.1053/meta.2002.32723. PMID 12037719
- [Background] Oliveira CLP, Boule NG, Berg A, Sharma AM, Elliott SA, Siervo M, Ghosh S, Prado CM. Consumption of a High-Protein Meal Replacement Leads to Higher Fat Oxidation, Suppression of Hunger, and Improved Metabolic Profile After an Exercise Session. Nutrients. 2021 Jan 5;13(1):155. doi: 10.3390/nu13010155. PMID 33466462
- [Background] Kendzierski, D., & DeCarlo, K. J. (1991). Physical Activity Enjoyment Scale: Two Validation Studies. Journal of Sport and Exercise Psychology, 13(1), 50-64. doi:10.1123/jsep.13.1.50.
- [Background] Rothschild JA, Kilding AE, Broome SC, Stewart T, Cronin JB, Plews DJ. Pre-Exercise Carbohydrate or Protein Ingestion Influences Substrate Oxidation but Not Performance or Hunger Compared with Cycling in the Fasted State. Nutrients. 2021 Apr 14;13(4):1291. doi: 10.3390/nu13041291. PMID 33919779